CLINICAL TRIAL: NCT06762392
Title: Effectiveness of Blood Flow Restriction in Postoperative Rehabilitation for Anterior Cruciate Ligament Injuries. A Pilot Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-3498956
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: Physical Therapy; Rehabilitation; Anterior Cruciate Ligament; Blood Flow Restriction; Randomized Clinical Trial
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Rehabilitation (Active Comparator): Participants in this group will receive a standardized post-operative rehabilitation protocol specifically designed for ACL reconstruction recovery. The protocol includes progressive exercises tailored to the recovery phases: early recovery (Phase 1), strength and neuromuscular control (Phase 2), agility and landing mechanics (Phase 3), and return to sport (Phase 4). Sessions will be supervised weekly by trained Physical Therapists, with additional unsupervised exercises to be performed at home or in the gym. This protocol follows current evidence-based guidelines without the incorporation of blood flow restriction therapy
  Interventions: Other: Standard Rehabilitation
- Standard Rehabilitation + Blood Flow Restriction (Experimental): Participants in this group will follow the same standardized post-operative rehabilitation protocol as the Active Comparator group, tailored to the recovery phases for ACL reconstruction (Phases 1-4). In addition, during Phase 2 (weeks 2-12), participants will undergo blood flow restriction (BFR) therapy during specific strengthening exercises. The BFR intervention involves applying a pneumatic cuff to the proximal thigh to achieve 70-80% arterial occlusion, combined with low-intensity resistance exercises (15-20% of 1RM). This approach aims to enhance muscle strength and recovery while minimizing joint stress. Sessions will be supervised weekly by trained Phyisical Therapists.
  Interventions: Other: Blood Flow Restriction

INTERVENTIONS:
Other: Blood Flow Restriction — Blood Flow Restriction (BFR) therapy in this study involves the application of a pneumatic cuff around the proximal thigh to restrict arterial blood flow during specific rehabilitation exercises. The cuff will be inflated to achieve 70-80% of arterial occlusion, while participants perform low-intensity resistance exercises at 15-20% of their one-repetition maximum (1RM). BFR therapy will be used during Phase 2 of rehabilitation (weeks 2-12) alongside a standardized rehabilitation protocol. The intervention will be closely monitored by trained Physical Therapists to ensure safety and efficacy, with pressure adjustments made in real-time based on the participant's exercise performance. This intervention distinguishes itself by its use of BFR, a technique that is not part of conventional ACL rehabilitation
  Arms: Standard Rehabilitation + Blood Flow Restriction
Other: Standard Rehabilitation — The Standard Rehabilitation (RHB) intervention in this study consists of a structured, evidence-based protocol designed to optimize recovery after anterior cruciate ligament (ACL) reconstruction. This rehabilitation protocol is implemented across four phases. The rehabilitation will be supervised by experienced Physical Therapists, and participants will be given a tailored home exercise program to complement the supervised sessions. The intervention aims to optimize recovery, restore function, and reduce the risk of re-injury.
  Arms: Standard Rehabilitation

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of adding Blood Flow Restriction (BFR) therapy to a standardized rehabilitation protocol in patients undergoing postoperative rehabilitation following anterior cruciate ligament (ACL) repair surgery.

The main questions it aims to answer are:

Does combining BFR therapy with a standardized rehabilitation protocol improve functional recovery compared to rehabilitation alone?

Does the addition of BFR therapy enhance muscle strength and reduce recovery time in patients after ACL repair surgery?

Participants will undergo their assigned rehabilitation protocol and will be assessed prior to and after the intervention to determine if the addition of BFR therapy to the standard rehabilitation programme significantly improves functional recovery, muscle strength, and overall rehabilitation outcomes following ACL repair surgery.

DETAILED DESCRIPTION:
Anterior Cruciate Ligament (ACL) reconstruction is a common surgical intervention following ligament rupture, particularly among athletes engaged in pivoting sports such as soccer, handball, volleyball, and skiing. Despite surgical advances, up to 35% of athletes fail to return to their pre-injury level within two years post-surgery, with factors such as fear of re-injury and neuromuscular deficits playing a significant role.

This randomized controlled trial evaluates the efficacy of integrating Blood Flow Restriction (BFR) therapy into standard rehabilitation protocols after ACL reconstruction. Participants aged 18-45 years, recovering from ACL surgery, will be randomized into two groups: a control group following the standard rehabilitation protocol and an experimental group combining BFR therapy with rehabilitation. BFR involves applying controlled vascular restriction to the proximal limb using automated devices during low-intensity resistance exercises, aiming to enhance strength and neuromuscular recovery safely.

The intervention spans 12 weeks, primarily focusing on the strength and neuromuscular control phase of rehabilitation. Outcomes will include measures of pain, fear of movement, functional performance, and readiness to return to sport. Evaluations will be conducted at baseline and at 2, 6 and 12 weeks post-surgery. The study seeks to determine whether BFR accelerates recovery, improves functional outcomes, and facilitates a safer, more effective return to athletic activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 45 years.
* Patients who have undergone anterior cruciate ligament (ACL) reconstruction surgery

Exclusion Criteria:

* Cardiovascular comorbidities
* Severe metabolic disorders or postoperative complications
* Previous joint disorders requiring surgery on the affected leg
* Pregnancy
* Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From baseline to the end of the intervention at 24 weeks
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a self-reported measure where the participant marks their perceived pain on a 100mm line, with one end representing "no pain" and the other representing the "worst pain imaginable." The VAS provides a subjective measure of pain intensity, enabling the tracking of pain levels over time to evaluate the impact of the intervention on pain relief. This is a commonly used tool to gauge pain perception in both clinical and research settings.
Strength | From baseline to the end of the intervention at 24 weeks
  Strength will be assessed using handheld dynamometry, an objective measure of muscle force production. Participants will perform maximal voluntary contractions against the dynamometer, which quantifies force output in Newtons (N) or kilograms (kg). This method provides a reliable and valid measure of muscle strength, allowing for the evaluation of changes over time in response to the intervention.
Range of Motion | From baseline to the end of the intervention at 24 weeks
  Range of Motion (ROM) will be assessed using goniometry, a standardized method for measuring joint flexibility and movement capacity. A goniometer will be positioned at the joint of interest, and participants will perform active and/or passive movements while the angular displacement is recorded in degrees. This technique provides an objective measure of joint mobility, enabling the evaluation of changes over time in response to the intervention

SECONDARY OUTCOMES:
Kinesiophobia | From baseline to the end of the intervention at 24 weeks
  Kinesiophobia, or the fear of movement due to pain or injury-related concerns, will be assessed using the Tampa Scale for Kinesiophobia-11 (TSK-11), a validated self-reported questionnaire. The TSK-11 consists of 11 items that evaluate fear-avoidance beliefs related to movement and physical activity. Participants rate their level of agreement with each statement on a Likert scale, generating a total score that reflects the severity of movement-related fear.
Patient's Quality of Life | From baseline to the end of the intervention at 24 weeks
  Quality of life will be assessed using the 12-Item Short Form Health Survey (SF-12), a validated self-reported questionnaire that measures physical and mental health status. The SF-12 evaluates key domains such as physical functioning, pain, general health perceptions, vitality, social functioning, emotional well-being, and mental health. Scores are calculated to generate composite measures of physical and mental health, allowing for the assessment of overall well-being and the impact of the intervention on participants' quality of life
Functional Performance | From baseline to the end of the intervention at 24 weeks
  Functional performance will be assessed through a series of validated physical tests designed to evaluate lower limb strength, endurance, and neuromuscular control. Participants will complete the following tests (1) Single Heel Rise (Step Test): The participant stands on one leg on a step and performs repeated heel raises until fatigue or failure to maintain proper form. This test assesses calf muscle endurance and strength (2) Single Leg Bridge: The participant lies supine with their heel positioned 60 cm above the floor and performs repeated single-leg hip bridges. This test evaluates posterior chain strength, particularly in the gluteal and hamstring muscles (3) Single Leg Squat: The participant performs a squat on one leg, aiming to reach 60° of knee flexion while maintaining balance and proper form. This test measures lower limb strength, stability, and motor control.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No